CLINICAL TRIAL: NCT05793138
Title: Integration of Geriatric Care Into Dialysis Clinics
Brief Title: Dialysis Geriatric Care Model
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00112850
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Diseases; Dialysis; Geriatric
Keywords: Dialysis; Quality of life; Care Model
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Placebo Comparator): Participants will receive usual dialysis care for 12 months, then they will receive the geriatric care model.
  Interventions: Behavioral: Usual Care
- Geriatric Care Model (Active Comparator): Participants will complete the GOLD, along with a few additional short surveys and a Short Physical Performance Battery. Information gathered will guide the research geriatric team's recommendation report to the participants' dialysis care team. The dialysis teams will receive training on how to use the recommendation report and local resources to initiate geriatric problem management. Participants will be seen every 4 months for follow-up for roughly 12 months.
  Interventions: Behavioral: Geriatric Care Model

INTERVENTIONS:
Behavioral: Geriatric Care Model — First, older adults complete the Geriatric screen for OLder adults receiving Dialysis (GOLD), a battery of validated, self-administered geriatric screening instruments, used to identify Geriatric 5M-related problems. Then, a research team with geriatrics expertise leads patient prioritization of GOLD-identified problems in a telehealth visit and provides the dialysis team with guideline-directed, individualized recommendations for geriatric problem management.
  Arms: Geriatric Care Model
Behavioral: Usual Care — Participants will continue to receive standard of care. Then after 12 months, they will follow the Geriatric Care Model. They will complete the Geriatric screen for OLder adults receiving Dialysis (GOLD), a battery of validated, self-administered geriatric screening instruments, used to identify Geriatric 5M-related problems. Then, a research team with geriatrics expertise leads patient prioritization of GOLD-identified problems in a telehealth visit and provides the dialysis team with guideline-directed, individualized recommendations for geriatric problem management.
  Arms: Usual Care

SUMMARY:
The objectives of this study are to refine the dialysis care model with key stakeholder input and conduct a pilot randomized controlled trial (RCT) to obtain evidence critical to inform a definitive RCT.

DETAILED DESCRIPTION:
The investigators designed a new dialysis care model that includes a centralized geriatric team that uses information from the Geriatric screen for OLder Dialysis patients (GOLD) to develop individualized recommendations for geriatric syndrome management based on the patient's priorities. The study population is older adults receiving hemodialysis and dialysis staff. The investigators will have patient participants complete the care model and undergo geriatric evaluation. This phase will be referred to as refinement aim 1. The investigators will then assess agreement of each GOLD instrument with its corresponding geriatric evaluation. The investigators will assess acceptability and feasibility of the care model through surveys and interviews with patients and dialysis staff to complete refinement aim 2. Once the new dialysis care model is redefined, the investigators will conduct the third phase, pilot RCT (geriatric care model vs. usual care) and assess geriatric problem management at 4 months, as well as, patient reported outcomes, physical function, and health care utilization at intervals up to 12 months. The analyses will include 1) measure of agreement using Cohen's kappa, 2) qualitative rapid analyses, 3) descriptive statistics from acceptability and feasibility surveys, 4) descriptive statistics from pilot RCT data, and 5) tests for difference in geriatric problem management between treatment and control groups. The study does not involve activity from participants that would exceed normal or routine care so there are negligible physical, financial, or legal risks.

ELIGIBILITY:
Patient Inclusion Criteria:

* community-dwelling dialysis patients 55 and older
* may have cognitive impairment

Patient Exclusion Criteria:

* advanced dementia
* non-English or Spanish speaking
* nursing home residents
* hospice enrollees

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in geriatric problem management as measured by survey | Baseline, 4, 8, 12 months
  Problems include depression, anxiety, difficulty with memory, difficulty with daily activities, falling or fear of falling, obtaining and following instructions for taking medications, having unwelcome side effects from medications, not having enough support from others, and not having access to or eating enough food. The score for each problem ranges from 0 to 4, where a higher score indicates better management of the problem.

SECONDARY OUTCOMES:
Practicality as measured by amount of time utilized by study personnel to conduct RCT (randomized controlled trial) | up to 12 months
Practicality as measured by number of resources utilized by study personnel to conduct RCT (randomized controlled trial) | up to 12 months
Fidelity as measured by number of completed study visits | up to 12 months
Retention as measured by number of participants who complete the study | up to 12 months
Recruitment as measured by number of participants enrolled | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rasheeda K Hall, MD, MBA, MHS, FASN, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No